CLINICAL TRIAL: NCT03774069
Title: Evaluation of Remote Consultation to Patients With Type 1 Diabetes Under Continuous Glucose Sensors and Insulin Pump Therapy Using the DreaMed Advisor Pro. An Open Label, Randomized Non-inferiority Study of Insulin Pump Therapy Adjustments Between DreaMed Advisor Pro and Standard of Care-The Advisor Pro Direct Study
Brief Title: The Advisor Pro Direct Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was finally decided not to perform the interventional part of the study. Only the questionnaire's part was performed
Sponsor: Rabin Medical Center (Other)
Collaborators: DreaMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC040818ctil
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Insulin pump treatment; Type 1 diabetes; Pump setting advisor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DreaMed Advisor Pro (Experimental): Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted using the DreaMed Advisor pro.
  Interventions: Device: DreaMed Advisor Pro
- Control group- medical guided recommendation (Active Comparator): Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ration and insulin activity time) will be adjusted by the medical team
  Interventions: Other: Medical guided recommendation

INTERVENTIONS:
Device: DreaMed Advisor Pro — Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted using the DreaMed Advisor Pro and sent directly to the patient
  Arms: DreaMed Advisor Pro
Other: Medical guided recommendation — Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted by the medical team according to standard of care
  Arms: Control group- medical guided recommendation

SUMMARY:
The DreaMed Advisor Pro is a software which automatically analyses treatment information, learns patient's needs and accordingly suggests adjustments in insulin dosing. DreaMed Advisor Pro is a decision- support software intended for assisting healthcare professionals in the management of type 1 diabetes patients who use insulin pumps as their insulin delivery therapy and monitor their blood glucose levels using CGM (Continuous Glucose Monitoring) or CGM and self-management blood glucose meter.

The main objective of the proposed study is to test the safety, reliability, and efficacy of the DreaMed Advisor Pro algorithm when the recommendation is sent directly to the patient without a physician review.

Participants will be randomized in a 1:1 ratio to either the intervention group (DreaMed Advisor Pro) or control group (standard of care). Participants will download the CGM and pump data at no less frequent than every 4 weeks for both groups during the 3 months period of the study.

Each time new data is received, the following actions will be performed:

In the intervention group, a new algorithm recommendation for pump settings will be issued. The recommendation will be approved by a technical, non-physician to assure that glucose data are not fall within predefined safety criteria which require a physician approval before the recommendation will be sent to the patient, otherwise, recommendation will be sent directly to the patient.

In the control group, if no safety criteria is met, it is the responsibility of the patient to contact his/her physician to advise on change of treatment. In case a safety issue has occurred, the physician will contact the patient and change the pump settings.

Prior to initiating the interventional phase of the study, we will evaluate the experience of patients in self adjustments of insulin dosing in regular care management and to evaluate their acceptance for using an automated dosing recommendations software. The evaluation will be done by asking patients/caregivers to fill 15 questions survey. 100 patients are anticipated to participate in this phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with type 1 diabetes (>1 yr diagnosis)
2. Age- 6-30 years old
3. HbA1c equals or above 7% and equals or below 10%
4. Insulin infusion pump CSII (Continuous Subcutaneous Inulin Infusion) therapy for at least 4 months and current treatment with one of the following pumps: Omnipod Insulet (Bedford, MA), Medtronic Minimed Veo insulinPump (MMT-754, MMT-554), Medtronic 640G or Animas.
5. BMI below 30 kg/m^2
6. Patients willing to follow study instructions (willing to measure capillary blood glucose as required by their glucose sensor for calibration and use the bolus- calculator feature of the pump)
7. Patients are required to have minimum computer skills and understanding of navigating the internet.
8. Patients are required to know basic English.
9. Patients willing to use glucose sensor for study duration.
10. Patients will have to have a smartphone (Apple or Android) or PC with email account.

Exclusion Criteria:

1. An episode of diabetic ketoacidosis within the month prior to study entry
2. Any significant diseases/ conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise patient's safety.
3. Current participation in any other interventional study.
4. Known or suspected allergy to trial products such as adhesives, tapes, needles.
5. Female subject who is pregnant or lactating or planning to become pregnant within the planned study duration
6. Severe hypoglycemia within six months prior to enrollment as defined by the ADA and Endocrine society as follows: Severe hypoglycaemia is an event requiring assistance of another person (due to change in mental status) to actively administer carbohydrates, glucagon, or take othe corrective actions.
7. Current use of the following medications: medications that are use to lower blood glucose such as Pramlintide, Metformin and GLP-1 analogs. Beta blockers, glucocorticoids and other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
8. Hypoglycemia unawareness
9. Relevant severe organ disorders (diabetic nephropathy, diabetic retinopathy, diabetic foot syndrome) or any secondary disease or complication of diabetes mellitus.

   * Subject has unstable or rapidly progressive renal disease or is receiving dialysis.
   * Subject has active proliferative retinopathy.
   * Active gastroparesis
10. Patient suffers from eating disorder. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage of glucose readings within range of 70-180 mg/dl (3.9 to 10mmol/L) | Final visit (week 12)
Percentage of readings below 54 mg/dl (3.3 mmol/l) | Final visit (week 12)

SECONDARY OUTCOMES:
HbA1c | Final visit (week 12)
Diabetes treatment satisfaction questionnaire | Final visit (week 12)
  The questionnaire contains 12-14 items (12 for the teens version and 14 for the parents version) the subscale for each items is from 0 to 6, and for most items the the higher the score, the greater the satisfaction with the treatment.Subscales are summed. More specific instruction for analysis are detailed in Diabetologia 52:(suppl 1) S397, Abstruct 1013 and in a document named "Summary of recommended scoring" by Prof. Bradley, University of London
Percentage of glucose readings below 70 mg/dl (3.9 mmol/L) | Final visit (week 12)
Percentage of readings below 60 mg/dl (3.35mmol/L) | Final visit (week 12)
Percentage of readings above 180 mg/dl (10.0mmol/L) | Final visit (week 12)
percentage of readings above 250 mg/dl (13.9 mmol/L) | Final visit (week 12)
Area above the curve of glucose level of 180 mg/dl | Final visit (week 12)
Area above the curve of glucose level above180 mg/dl | Final visit (week 12)
Area under the curve of glucose level of 70 mg/dl | Final visit (week 12)
Area under the curve of glucose level below 70 mg/dl | Final visit (week 12)
Mean sensor blood glucose | Final visit (week 12)
Glucose variability measured by standard deviation | Final visit (week 12)
Number of recommendations sent to patient in the last 6 months prior to baseline and during intervention period | Final visit (week 12)
Number of recommendations for changes in settings per patient | Final visit (week 12)
Number of recommendations for changes in settings per iteration | Final visit (week 12)
Number of physician override Advisor recommendation | Final visit (week 12)

CONTACTS AND LOCATIONS:
Locations (1):
- Schnider Children's medical center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No